CLINICAL TRIAL: NCT05283902
Title: Effectiveness, Immunogenicity and Safety of the Second Booster Dose (Fourth Dose) of the Vaccine Against COVID-19 in the Elderly: Study Reforça Mais (Plus Booster)
Brief Title: Effectiveness, Immunogenicity and Safety of the Second Booster Dose of the Vaccine Against COVID-19 in the Elderly
Acronym: Plus_Booster
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Federal University of Espirito Santo (Other)
Collaborators: Secretaria de Estado da Saúde do Espírito Santo - SESA (Unknown); Centro de Pesquisas René Rachou (Other Government)
Responsible Party: Principal Investigator, Valéria Valim, Professor, Federal University of Espirito Santo
Other Study IDs: FUES05
Record Dates: First submitted 2022-03-10; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Vaccine Adverse Reaction; Vaccine-Preventable Diseases
MeSH Terms: conditions — COVID-19; Vaccine-Preventable Diseases | interventions — ChAdOx1 nCoV-19; BNT162 Vaccine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (cellular and humoral immune response)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Effectiveness group: There are an estimated 490,000 eligible individuals aged 60 and over statewide for the effectiveness study.
  Interventions: Biological: ChAdOx1 nCoV-19 or Comirnaty or Janssen COVID-19 Vaccine
- Elderly group - Immunogenicity: 240 participants from the Effectiveness group, with quotas distributed by sex (50% male and 50% female) and age group, will be invited to participate in biological sample collection for the immunogenicity study.
  Interventions: Biological: ChAdOx1 nCoV-19 or Comirnaty or Janssen COVID-19 Vaccine
- Immunosupressed group: 240 biorepository samples from a cohort of immunosuppressed patients with autoimmune diseases who received the fourth dose, in a study conducted by the same team of researchers.
  Interventions: Biological: ChAdOx1 nCoV-19 or Comirnaty or Janssen COVID-19 Vaccine

INTERVENTIONS:
Biological: ChAdOx1 nCoV-19 or Comirnaty or Janssen COVID-19 Vaccine — In a Technical Note, the State of Espírito Santo decided to recommend the application of the fourth dose with vaccines using messenger RNA (mRNA) technology or viral vector vaccine, for all people aged 60 years or older, with an interval of 90 days from of the third dose, considering that, while there is no availability of vaccines adapted to the new variants, boosters with available vaccines are still the most appropriate ways to prevent hospitalization and deaths.

SUMMARY:
The objective of this observational case-crossover study is to evaluate the effectiveness, safety and immunogenicity of the second booster dose in the elderly. There are an estimated 490,000 eligible individuals aged 60 and over statewide for the effectiveness study. Two hundred and forty participants will be invited to participate in biological sample for the immunogenicity study. This sub-sample will be compared with 240 biorepository samples from a cohort of immunosuppressed patients with autoimmune diseases who received the fourth dose, in a study conducted by the same team of researchers. The main effectiveness outcome will be the number of hospitalizations; and secondary outcomes will be deaths, number of reported cases, number of cases confirmed by RT-PCR. The safety assessment will be carried out by monitoring adverse events. The cellular and humoral immune response will be evaluated by viral neutralization assay (search for neutralizing antibodies), serological assay by chemiluminescence, determination of specific IgM and IgG profile, dosage of soluble systemic factors (chemokines, cytokines and growth factors), stimulation in vitro antigen-specific peripheral blood mononuclear cells and investigation of memory T and B lymphocytes and intracytoplasmic cytokines. The study hypothesis is that elderly people who received the second booster dose have a lower incidence rate of hospitalizations and death than those who received the primary regimen (two doses or one of Janssen) or a booster dose, and that the immune response humoral and cellular function of the elderly is similar to those who are immunosuppressed.

DETAILED DESCRIPTION:
Faced with the new scenario of high transmission of the Ômicron variant of SARS-COV-2, in which the elderly over 60 years and immunosuppressed even vaccinated with three doses have become a population vulnerable to a greater probability of serious illness by Covid-19, demanding an increase in risk of hospitalization and deaths, the application of the fourth dose (second booster dose) has become an alternative to increase protection for these individuals. The general objective of this study is to evaluate the effectiveness, safety and immunogenicity of the second booster dose in the elderly. This is an observational, case-crossover study, based on databases with notification and vaccination records and a cohort study for the analysis of immunogenicity. Elderly people of both sexes aged 60 years or older, residents of Espírito Santo, will be included. There are an estimated 490,000 eligible individuals aged 60 and over statewide for the effectiveness study. Two hundred and forty participants, with quotas distributed by sex (50% male and 50% female) and age group, will be invited to participate in biological sample collection on the day of application of the second booster dose (T1) , 28 days after the second booster dose (T2), at the follow-up visit after 3 months (T3), 150 days (T4) and 180 days (T5), for follow-up of vaccine response and follow-up of duration of immunity, in a health unit in Cariacica-ES. This sub-sample will be compared with 240 biorepository samples from a cohort of immunosuppressed patients with autoimmune diseases who received the fourth dose, in a study conducted by the same team of researchers. The main effectiveness outcome will be the number of hospitalizations, weighted by protection time, 90 days after complete immunization (14th day after second booster dose); and secondary outcomes will be deaths, number of reported cases, number of cases confirmed by RT-PCR. The safety assessment will be carried out by monitoring adverse events. The cellular and humoral immune response will be evaluated by viral neutralization assay (search for neutralizing antibodies), serological assay by chemiluminescence, determination of specific IgM and IgG profile, dosage of soluble systemic factors (chemokines, cytokines and growth factors), stimulation in vitro antigen-specific peripheral blood mononuclear cells and investigation of memory T and B lymphocytes and intracytoplasmic cytokines. The study hypothesis is that elderly people who received the second booster dose have a lower incidence rate of hospitalizations and death than those who received the primary regimen (two doses or one of Janssen) or a booster dose, and that the immune response humoral and cellular function of the elderly is similar to those who are immunosuppressed.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 60 years
* Residents of Espírito Santo, Brazil

Exclusion Criteria:

* Being under active treatment (chemotherapy and/or radiotherapy) for the treatment of any type of neoplasm
* Being admitted to an institutionalization establishment for the elderly (hospitals, nursing homes, shelters or similar).
* Patients with mental illness with inability to understand the consent form

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are an estimated 490,000 eligible individuals aged 60 and over statewide for the effectiveness study. Two hundred and forty participants, with quotas distributed by sex (50% male and 50% female) and age group, will be invited to participate in biological sample collection for the immunogenicity study, in a health unit in Cariacica-ES. This sub-sample will be compared with 240 biorepository samples from a cohort of immunosuppressed patients with autoimmune diseases who received the fourth dose, in a study conducted by the same team of researchers.
Sampling Method: Non-Probability Sample
Enrollment: 490000 (Estimated)
Dates: Start 2022-03-19 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
number of hospital admissions | Change from baseline at 6 months
  number of hospital admissions for covid-19 recorded in the "e-SUS notifica"
Number of adverse events | Change from baseline at 1 month
  Surveillance of adverse post-vaccine events (PVAE) and adverse events of special interest (EAIE) recorded in the "e-SUS notifica"

SECONDARY OUTCOMES:
number of deaths | Change from baseline at 6 months
  Number of deaths with specific ICD for covid-19 recorded in the "e-SUS notifica"
number of Covid-19 cases | Change from baseline at 6 monhts
  number of Covid-19 cases confirmed by RT-PCR recorded in the "e-SUS notifica"
Viral neutralization assay | Change from baseline at 1, 3, 5 and 6 months
  Neutralizing antibody titers will be expressed by the ability of antibodies to neutralize up to 50% the number of plaques (PRNT50). Title > 1:50 will be considered positive.
Serological assay | Change from baseline at 1, 3, 5 and 6 months
  Serological test by chemiluminescence for qualitative and quantitative determination of specific IgG antibodies against the nucleocapsid protein of SARS-Cov-2. Results are expressed in U/mL and data interpretation will be done as follows: <0.8 U/mL = non-reactive sample; ≥0.8 U/mL = reactive sample.
Soluble systemic factors | Change from baseline at 1, 3, 5 and 6 months
  Dosage of soluble systemic factors (chemokines, cytokines and growth factors). Results will be expressed in pg/ml.
Lymphocyte investigation | Change from baseline at 1, 3, 5 and 6 months
  Investigation of memory T and B lymphocytes. The results will be expressed in percentage positive frequency for a specific cell phenotype.
Cytokine investigation | Change from baseline at 1, 3, 5 and 6 months
  Investigation of intracytoplasmic cytokines. The results will be expressed in percentage positive frequency for a specific cell phenotype.

CONTACTS AND LOCATIONS:
Locations (1):
- Valéria Valim, Vitória, Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: No